CLINICAL TRIAL: NCT06891027
Title: Loss of Parental Workforce in Paediatric Fractures
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Berkay Girgin, Principal Investigtor, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2024-1169
Record Dates: First submitted 2025-03-14; First posted 2025-03-24 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Fractures; Lower Extremity Fractures; Upper Extremity Fractures
Keywords: pediatric fracture; parental workforce; loss of workforce

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- pediatric fracture: all paediatric (<18 years) patients presenting with a fracture will be included in the study. parents of patients presenting with a fracture will be informed about the study and parents who are willing to participate in the study will be included. parents will be given a form indicating various workforce losses (including housework and social life) at the first application. this form will be received from the parents at the end of treatment. study data will be collected on this form.

SUMMARY:
Childhood fractures are frequently encountered in orthopaedic practice. 40-64% of boys and 25-40% of girls have at least one fracture by the age of 16. Children, who are more fragile than adults, usually require additional care support during the treatment process. Labour force statistics have determined that one third of the loss of labour force occurs after musculoskeletal injuries.

When the literature is examined, there are many studies investigating loss of labour force after fractures. It was found that 20% of the patients never returned to work after distal radius fracture and the average loss of labour force was 9.2 weeks. In another study, while the return to work period was 60 days in minor hand injuries, it was reported that the return to work could increase to 360 days in major hand injuries. In another study, the average return to work time in patients aged >50 years with fragility fractures was found to be 20.5 days. The rate of return to work after traumatic spinal fracture was found to be only 38.1%.

In daily practice, the investigators observe that parents frequently do not go to work for child care after child fractures. However, there is no similar study investigating this loss of labour force after pediatric fractures in the literature. In this study, the investigators aimed to investigate the loss of parental labour force (LWL) in conservatively followed pediatric fractures

ELIGIBILITY:
Inclusion Criteria:

* patients <18 years of age who underwent plaster splinting for any extremity fracture

Exclusion Criteria:

* Parents of patients aged >18 years
* Parents of patients undergoing surgical treatment
* Parents of patients whose initial diagnosis or follow-up was performed at an external centre
* Patients with one parent not working (patients with one working parent will be excluded)
* Parents of patients who did not want to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Parents of patients aged <18 years who were admitted to Ankara Etlik City Hospital Emergency Orthopaedics and Traumatology Outpatient Clinic and other Orthopaedics and Traumatology Outpatient Clinics and underwent plaster splinting due to any extremity fracture
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Loss of Parental Workforce Questionnaire | from first presentation after fracture to the end of treatment (approximately 6 weeks in conservative cases, 3 months in surgical treatments)
  A questionnaire called "Loss of Parental Workforce Questionnaire" will be used to evaluate the parental workforce loss. Also with this questionnaire the effect of treatment choice (conservative or surgical) to parental workforce loss will be assessed.

SECONDARY OUTCOMES:
Children's Return to School Time | from first presentation after fracture to the end of treatment (approximately 6 weeks in conservative cases, 3 months in surgical treatments)
  "Loss of Parental Workforce Questionnaire" will also be used to assess Children's Return to School Time.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes